CLINICAL TRIAL: NCT02701296
Title: Assessment of Knee Pain in Patients Receiving Continuous Femoral Nerve Block Combined With Either Ultrasound Guided Posterior Capsular Injection or Selective Tibial Nerve Block Following Total Knee Arthroplasty
Brief Title: Posterior Capsular Injection With Femoral Nerve Block for Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trinity Health Of New England (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-10-004
Record Dates: First submitted 2016-02-17; First posted 2016-03-08 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Posterior Knee Infiltration
Keywords: Infiltration between popliteal artery and capsule of knee (iPACK)
MeSH Terms: interventions — Ropivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Posterior capsular injection (Experimental): Ultrasound guided posterior capsular injection of ropivacaine with epinephrine
  Interventions: Drug: Ropivacaine with Epinephrine
- Tibial nerve block (Active Comparator): Ultrasound selective tibial nerve block of ropivacaine
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine with Epinephrine — Posterior capsular injection - ultrasound guided infiltration of Ropivacaine with Epinephrine between popliteal artery and capsule of knee above the femoral condyles
  Other Names: Naropin; Adrenalin
  Arms: Posterior capsular injection
Drug: Ropivacaine — Tibial nerve block - ultrasound selective Ropivacaine tibial nerve block in the popliteal fossa
  Other Names: Naropin
  Arms: Tibial nerve block

SUMMARY:
To assess pain control after total knee replacement surgery using two different nerve block techniques. The 2 methods are:

1. Continuous femoral nerve block with ultrasound guided posterior capsular injection
2. Continuous femoral nerve block with ultrasound selective tibial nerve block.

DETAILED DESCRIPTION:
Patients undergoing total knee replacement surgery experience severe post-operative pain. Continuous femoral nerve block combined with selective tibial nerve block provides optimal pain control in the anterior and posterior aspect of the knee respectively. However, in patients with pre-existing neuropathy of the sciatic nerve, the blockade of tibial nerve is contraindicated because of increased risk of nerve damage that may lead to exacerbation of neurologic symptoms. In such patients where selective tibial nerve block cannot be offered, ultrasound guided posterior knee capsular injection may be an alternative technique for controlling posterior knee pain after surgery. Posterior capsular injection by surgeons intraoperatively, when combined with femoral nerve block has been shown to provide pain control after total knee replacement. With posterior capsular injection, the main trunk of the tibial nerve is spared and only the terminal nerve endings innervating the posterior knee joint is blocked providing effective pain control. In this study, the efficacy of ultrasound guided posterior capsular injections performed pre-operatively will be compared to tibial nerve block in controlling knee pain after surgery.

The results of this study may help establish the efficacy of ultrasound guided posterior capsular injection as an alternative to tibial nerve block in patients undergoing total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients having primary, unilateral total knee arthroplasty
* Age 18-80

Exclusion Criteria:

* History of neurologic disease, neuropathy, diabetes, or major systemic illness
* Allergy to local anesthetic solution or NSAIDs
* Pregnancy
* Chronic use of narcotics
* Inability to give consent/cooperate with study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-11-07 (Actual); Primary Completion 2014-08-31 (Actual); Study Completion 2014-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Sinha, Principal Investigator — Saint Francis Hospital and Medical Center
Locations (1):
- Saint Francis Hospital and Medical Center, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Posterior Capsular Injection | Tibial Nerve Block
Started | 42 | 38
Completed | 42 | 36 (Data was incomplete for two participants their data was not included in the overall data analysis.)
Not Completed | 0 | 2
Not completed — Incomplete Data | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Posterior Capsular Injection | Tibial Nerve Block | Total
Number analyzed (Participants) | 42 | 36 | 78
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.9 (8.0) | 63.5 (8.9) | 64.8 (8.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 19 | 43
  Male | 18 | 17 | 35
Region of Enrollment [Number; unit: participants]
  United States | 42 | 36 | 78

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity
Description: Mean Numeric Pain Rating Scale (NPRS) self-reported pain Intensity on a 11-point score (0=no pain to 10= worst possible) in Post Anesthesia Care Unit (PACU) and every 6 hours for 48 hours post surgery
Time Frame: 48 hours post surgery
Measure: Mean (Standard Deviation); unit: pain score
Arm/Group | Posterior Capsular Injection | Tibial Nerve Block
Number analyzed (Participants) | 42 | 36
pain score
  PACU Admission | 3.5 (2.95) | 3.2 (3.67)
  PACU Discharge | 2.1 (1.78) | 1.5 (1.73)
  6th hour | 1.9 (1.85) | 2.0 (2.17)
  12th hour | 2.0 (2.36) | 1.2 (2.03)
  18th hour | 2.3 (2.21) | 3.2 (2.36)
  24th hour | 2.7 (2.21) | 3.4 (2.42)
  30th hour | 2.6 (2.40) | 3.0 (2.43)
  36th hour | 2.5 (2.46) | 2.7 (2.53)
  42nd hour | 3.2 (1.82) | 3.2 (2.5)
  48th hour | 2.5 (1.98) | 3.4 (2.4)

2. Secondary Outcome: Opioid Consumption
Description: Amount of opioid used for the first 24 hours post surgery
Time Frame: 24 hours post surgery
Population: Mean consumption of Hydromorphone(mg) post-op day 1
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Posterior Capsular Injection | Tibial Nerve Block
Number analyzed (Participants) | 42 | 36
mg | 0.33 (0.655) | 0.42 (0.706)

3. Secondary Outcome: Plantar Flexion in the Tibial Nerve Distribution
Description: Blinded nurse assessment on a 3-point scale 0= normal (No Motor Block), 1= weak (Partial Motor Block), 2 = absent (Complete Motor Block)
Time Frame: Upon emergence from anesthesia in the PACU
Measure: Count of Participants; unit: Participants
Arm/Group | Posterior Capsular Injection | Tibial Nerve Block
Number analyzed (Participants) | 42 | 36
Participants
  Complete Motor Block | 1 | 0
  Partial Motor Block | 3 | 25
  No Motor Block | 38 | 11

4. Secondary Outcome: Cold Sensation in the Tibial Nerve Distribution
Description: Number of participants with a self reported on a 3-point scale; 0=normal (No Sensory Block), 1= absent cold perception but touch sensation in tact (Partial Sensory Block), 2= absence of touch sensation (Complete Sensory Block)
Time Frame: Upon emergence from anesthesia in the PACU
Measure: Count of Participants; unit: Participants
Arm/Group | Posterior Capsular Injection | Tibial Nerve Block
Number analyzed (Participants) | 42 | 36
Participants
  Complete Sensory Block | 1 | 6
  Partial Sensory Block | 7 | 27
  No Sensory Block | 34 | 3

5. Secondary Outcome: Dorsiflexion in the Peroneal Nerve Distribution
Description: Number of participants with a blinded nurse assessment on a 3-point scale 0= normal (No Motor Block), 1= weak (Partial Motor Block), 2 = absent (Complete Motor Block)
Time Frame: Upon emergence from anesthesia in the PACU
Measure: Count of Participants; unit: Participants
Arm/Group | Posterior Capsular Injection | Tibial Nerve Block
Number analyzed (Participants) | 42 | 36
Participants
  Complete Motor Block | 0 | 0
  Partial Motor Block | 1 | 4
  No Motor Block | 41 | 32

6. Secondary Outcome: Sensation in the Peroneal Nerve Distribution
Description: Number of participants with self reported on a 3-point scale; 0=normal (No Sensory Block), 1= absent cold perception but touch sensation in tact (Partial Sensory Block), 2= absence of touch sensation (Complete Sensory Block)
Time Frame: Upon emergence from anesthesia in the PACU
Measure: Count of Participants; unit: Participants
Arm/Group | Posterior Capsular Injection | Tibial Nerve Block
Number analyzed (Participants) | 42 | 36
Participants
  Complete Sensory Block | 2 | 1
  Partial Sensory Block | 3 | 11
  No Sensory Block | 37 | 24

ADVERSE EVENTS:
Time Frame: 24 hours after total knee replacement surgery
Arm/Group | Posterior Capsular Injection | Tibial Nerve Block
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/36
Other Adverse Events (participants affected / at risk) | 0/42 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No